CLINICAL TRIAL: NCT05654467
Title: A Phase 2, Randomized, Observer-Blind, Controlled, Age De-escalation, Dosage Escalation Study to Assess the Safety and Immunogenicity of a Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine in Healthy Young Children, Infants, and Neonates in Panama
Brief Title: Study of a Novel Type 3 Oral Poliomyelitis Vaccine in Panama
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); PT Bio Farma (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency); Technical Resources International, Inc. (TRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 101; U1111-1285-1905 (Other: WHO)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Poliomyelitis
Keywords: Vaccine tolerability; Vaccine safety; Vaccine reactogenicity; Vaccine viral shedding; Vaccine immunogenicity
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: A 12-arm, randomized, observer-blind, controlled, age de-escalation, dosage escalation study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Group 1: Young Children, nOPV3 10^5.5 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV3 at a dose level of 10^5.5 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Group 3: Young Children, nOPV3 10^6.0 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV3 at a dose level of 10^6.0 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Group 5: Young Children, nOPV3 10^6.5 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV3 at a dose level of 10^6.5 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Groups 2, 4 and 6: Young Children, mOPV3 (Active Comparator): 48 young children aged 1 to <5 years will receive 2 doses of mOPV3 at a dose level of ≥ 10^5.8 CCID50 on Day 1 and Day 29
  Interventions: Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)
- Group 7: Infants, nOPV3 10^5.5 CCID50 (Experimental): 240 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV3 at a dose level of 10^5.5 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)
- Group 9: Infants, nOPV3 10^5.5 CCID50 (Experimental): 240 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV3 at a dose level of 10^6.0 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)
- Group 11: Infants, nOPV3 10^6.5 CCID50 (Experimental): 140 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV3 at a dose level of 10^6.5 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)
- Groups 8, 10 and 12: Infants, mOPV3 (Active Comparator): 240 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of mOPV3 at a dose level of ≥ 10^5.8 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)
- Group 13: Neonates, nOPV3 10^5.5 CCID50 (Experimental): 120 neonates (day of birth + 3 days) will receive 2 doses of nOPV3 at a dose level of 10^5.5 CCID50 on Day 1 and Day 29.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Group 15: Neonates, nOPV3 10^6.0 CCID50 (Experimental): 120 neonates (day of birth + 3 days) will receive 2 doses of nOPV3 at a dose level of 10^6.0 CCID50 on Day 1 and Day 29.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Group 17: Neonates, nOPV3 10^6.5 CCID50 (Experimental): 120 neonates (day of birth + 3 days) will receive 2 doses of nOPV3 at a dose level of 10^6.5 CCID50 on Day 1 and Day 29.
  Interventions: Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3)
- Groups 14, 16 and 18: Neonates, mOPV (Active Comparator): 120 neonates (day of birth + 3 days) will receive 2 doses of mOPV3 at a dose level of ≥ 10^5.8 CCID50 on Day 1 and Day 29
  Interventions: Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3)

INTERVENTIONS:
Biological: Novel Live Attenuated Type 3 Oral Poliomyelitis Vaccine (nOPV3) — The nOPV3 vaccine containing approximately 10^5.5, 10^6.0, or 10^6.5 CCID50 per dose.
  Arms: Group 11: Infants, nOPV3 10^6.5 CCID50; Group 13: Neonates, nOPV3 10^5.5 CCID50; Group 15: Neonates, nOPV3 10^6.0 CCID50; Group 17: Neonates, nOPV3 10^6.5 CCID50; Group 1: Young Children, nOPV3 10^5.5 CCID50; Group 3: Young Children, nOPV3 10^6.0 CCID50; Group 5: Young Children, nOPV3 10^6.5 CCID50; Group 7: Infants, nOPV3 10^5.5 CCID50; Group 9: Infants, nOPV3 10^5.5 CCID50
Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 (mOPV3) — The Sabin Monovalent Oral Poliomyelitis Vaccine Type 3 control and challenge vaccine (mOPV3) containing ≥ 10^5.8 CCID50 per dose.
  Arms: Group 11: Infants, nOPV3 10^6.5 CCID50; Group 7: Infants, nOPV3 10^5.5 CCID50; Group 9: Infants, nOPV3 10^5.5 CCID50; Groups 14, 16 and 18: Neonates, mOPV; Groups 2, 4 and 6: Young Children, mOPV3; Groups 8, 10 and 12: Infants, mOPV3

SUMMARY:
The purpose of this clinical trial is to assess the safety and tolerability (primary objective), immunogenicity (primary and secondary objectives), fecal shedding of vaccine viruses (secondary objective) and the potential for neurovirulence of shed virus (secondary objective) of a novel oral polio type 3 vaccine, nOPV3, as compared to Sabin monovalent type 3 vaccine controls (mOPV3), in healthy young children (192 subjects), infants (860 subjects), and neonates (480 subjects).

DETAILED DESCRIPTION:
This multicentered, 12-arm phase 2 study will be the first pediatric evaluation of nOPV3 in healthy young children, infants, and newborns. This trial will be initiated once results in the adult phase 1 study of nOPV3 indicate that there are no safety concerns, and that the vaccine elicits demonstrable immunogenicity. Additionally, prior to enrolling into cohort 2, the adult phase 1 data must show no concerning signals of reversion of attenuating sites from a subset of Next Generation Sequencing.

This study is intended to provide critical data on safety, immunogenicity, and genetic stability, as well as to demonstrate the vaccine's ability to reduce fecal shedding following a challenge with the Sabin type 3 strain.

Enrollment in this pediatric study will be staggered into three age-descending cohorts of 6 treatment groups of escalated target dose levels for the nOPV3 vaccine: cohort 1 composed of 192 healthy young children 1 to <5 years of age who have completed their full routine polio immunization series; cohort 2 composed of 860 healthy infants 6 weeks of age not previously vaccinated (OPV/IPV) who will be primed with a dose of inactivated poliomyelitis vaccine (IPV) prior to OPV3 vaccination [a subset, of the infants (n=360) will also receive the challenge virus]; and cohort 3, composed of 480 healthy poliomyelitis unvaccinated neonates (day of birth +3 days).

Progression into the next cohort and groups within cohorts will depend on safety evaluations of the prior Phase 1 adult trial and Day 8 safety evaluation of the previous groups in prior cohorts in the study.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria for all participants:

1. Healthy, as defined by the absence of any clinically significant medical condition or congenital anomaly as determined by medical history, physical examination, and clinical assessment of the investigator.
2. Parent(s) or guardian(s) willing and able to provide written informed consent prior to performance of any study-specific procedure.
3. Resides in study area and parent(s) or guardian(s) understands and is able and willing to adhere to all study visits and procedures (as evidenced by a signed informed consent form [ICF] and assessment by the investigator).
4. Parent(s) or guardian(s) agrees for participant to receive all routine infant and childhood immunizations as per the approved protocol adjusted schedule.

Inclusion Criteria for cohort 1 participants only:

1. Male or female child from ≥1 to <5 years-of-age at the time of initial study vaccination.
2. Based on available documentation or parental/guardian(s) report, previously completed the primary poliomyelitis immunization series for the jurisdiction, with last dose received more than 28 days prior to initial study vaccination.

Inclusion Criteria for cohort 2 participants only:

1. Male or female infant expected to be 6 weeks of age (43rd to 49th day of life [with day of birth being the first day of life], inclusive + 6 day window), at the time of initial study vaccination.
2. Prior to study vaccination has received no doses of IPV or OPV, based on no evidence of such vaccination per available parental/guardian(s) report or documentation.

Inclusion Criteria for Cohort 3 participants only:

1. Male or female newborn (1st day of life + 3-day window), at the time of initial study vaccination.
2. Prior to study vaccination has received no doses of IPV or OPV vaccine, based on no evidence of such vaccination per available parental/guardian(s) report or documentation.

Exclusion Criteria

Exclusion Criteria for all participants:

1. For all participants the presence of anyone under 10 years of age in the participant's household (living in the same house or apartment unit) who does not have complete "age appropriate" vaccination status with respect to poliovirus vaccines at the time of study vaccine administration. For household members younger than 10 years of age appropriate vaccination is complete series of the primary poliomyelitis immunization series for the jurisdiction.
2. For all participants having a member of the participant's household (living in the same house or apartment unit) who has received OPV based on the vaccination records in the previous three months before study vaccine administration.
3. Any participating children attending day care or pre-school during their participation in the study until one month after their last study vaccine administration.
4. Moderate or severe (grade ≥ 2) acute illness at the time of enrollment/first study vaccination-temporary exclusion (see Appendix II: Severity Grading Tables). Participant with mild (grade 1) acute illnesses may be enrolled at the discretion of the investigator.
5. Presence of fever on the day of enrollment/first study vaccination (axillary temperature

   ≥37.5˚C)-(Temporary exclusion for cohorts 1 and 2). If resolved in 48 hrs., can be enrolled.
6. A known allergy, hypersensitivity, or intolerance to any components of the study vaccines, including all macrolide and aminoglycoside antibiotics (e.g., erythromycin and kanamycin).
7. Any self-reported known or suspected immunosuppressive or immunodeficiency condition (including HIV infection) in the participant or household member (living under the same roof/in the same building rather than in the same compound).
8. Receipt of any systemic immune-modifying or immunosuppressant drugs prior to the first study vaccine dose or planned use during the study of study participants or a household member.
9. Any known or suspected bleeding disorder in the participant that would pose a risk to venipuncture or intramuscular injection.
10. Presence of severe malnutrition (weight-for-length/height z-score ≤-3SD median [per WHO published child growth standards])-temporary exclusion if marginal and subsequently gains weight.
11. Participation in another investigational product (drug or vaccine) clinical trial within 30 days prior to entry in this study or receipt of any such investigational product other than the study vaccine within 30 days prior to the first administration of study vaccine, or planned use during the study period.
12. Receipt of transfusion of any blood product or immunoglobulins within 12 months prior to the first administration of study vaccine or planned use during the study period.
13. Parent(s) or guardian(s) or participant has any condition that in the opinion of the investigator would increase the participant's health risks in study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments).

Exclusion Criteria for cohort 2 and 3 participants only:

1. Premature birth (less than 37 weeks gestation or less than 2500 grams birth weight).
2. From multiple birth (due to increased risk of OPV transmissions between siblings).

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1532 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious adverse events (SAEs) | Up to last visit for last subject, around 18 months
  Serious adverse event is any adverse event that results in any of the following outcomes:
  1. Death
  2. Is life-threatening (life-threatening means that the study participant was, in the opinion of the site PIs or PATH, at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).
  3. Requires inpatient hospitalization or prolongation of existing hospitalization.
  4. Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  5. Congenital abnormality or birth defect.
  6. Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant and require medical or surgical intervention to prevent one of the outcomes listed in the above definition of serious adverse event.
Frequency of solicited adverse events (AEs) for 7 days (day of vaccination and 6 following days) after each vaccination | Vaccination to 7 days post vaccination
  Solicited AEs are pre-specific AEs that are common or known to be associated with vaccination that are actively monitored as potential indicators of vaccine reactogenicity.
  The following specific solicited AEs will be monitored for this trial:
  Fever (axillary temperature ≥ 37.5°C) Vomiting Diarrhea Irritability Decreased feeding or appetite Fatigue or decreased activity
Frequency of unsolicited AEs for 28 days (day of vaccination and 27 following days) after each vaccination | From vaccination to 28 days post vaccination
  Unsolicited AEs are any AEs reported spontaneously by the participant's parent, observed by the study personnel during study visits or identified during review of medical records or source documents. In the absence of a diagnosis, abnormal physical examination findings or abnormal clinical safety laboratory test results that are assessed by the investigator to be clinically significant will be reported as an AE.
Post-vaccination frequency of seroconversion of type 3 anti-polio serum neutralizing antibody (NAb) in infants. | 28 days post second vaccination
  For previously vaccinated cohorts, seroconversion will be defined as a minimum 4-fold rise in titer relative to the baseline value among those initially seropositive.

SECONDARY OUTCOMES:
Post-vaccination frequency of seroconversion of type 3 anti-polio serum NAb | Baseline and 28 days post vaccination (Day 1 and Day 29 for neonates; Day 29,Day 57 and Day 85 for infants; Day 1, Day 29 and Day 57 young children)
  For previously vaccinated cohorts, seroconversion will be defined as a minimum 4-fold rise in titer relative to the baseline value among those initially seropositive and for unvaccinated neonates, seroconversion will be defined as a minimum 4-fold higher antibody titer relative to the expected level of maternal antibody.
Median type 3 anti-polio serum NAb titers | Baseline and 28 days post vaccination (Day 1, Day 29 and Day 57 for young children and neonates; Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV3, compared to that of mOPV3, following one or two doses in healthy young children, infants, and neonates.
Type 3 anti-polio serum NAb Geometric Mean Titer (GMT) | Baseline and 28 days post vaccination (Day 1, Day 29 and Day 57 for young children and neonates;Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV3, compared to that of mOPV3, following one or two doses in healthy young children, infants, and neonates.
Post-vaccination GMT ratios of type 3 anti-polio serum NAb, adjusted for baseline immunity | Baseline and 28 days post vaccination (Day 1, Day 29 and Day 57 for young children and neonates; Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV3, compared to that of mOPV3, following one or two doses in healthy young children, infants, and neonates.
Seroprotection rate, defined as type 3 anti-polio serum NAb reciprocal titer ≥ 8 | Baseline and 28 days post vaccination (Day 1, Day 29 and Day 57 for young children and neonates; Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV3, compared to that of mOPV3, following one or two doses in healthy young children, infants, and neonates.
Geometric mean fold rise (GMFR) in NAb titer relative to baseline for post-dose-1 and relative to post-dose-1 for post-dose-2. | Baseline and 28 days postvaccination (Day 1, Day 29 and Day 57 for young children and neonates; Day 29, Day57 and Day 85 for infants)
  Elicited by nOPV3, compared to that of mOPV3, in healthy young children, infants,and neonates.
Proportion of participants shedding type 3 poliovirus at any and at each post-vaccination stool collection, as assessed by polymerase chain reaction (PCR) in infants | Baseline through to 28 days post initial vaccination (Day 29 through to Day 57 for infants)
  After the initial dose of nOPV3, compared to mOPV3
Proportion of participants shedding type 3 poliovirus at any and at each post-challenge stool collection, as assessed by PCR in infants | Day of challenge through to 28 days post challenge (Day 113 through to Day 141, for infants)
  In participants negative for type 3 poliovirus in their last pre-challenge stool sample
Neurovirulence of shed study vaccine virus from select stool samples as measured by a transgenic mouse neurovirulence test in a subset of infants | Baseline through to 28 days post initial vaccination (Day 1 through to Day 29 for neonates)
  Within 28 days of an initial nOPV dose and compared to that of mOPV3

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Saez-Llorens, MD, Principal Investigator — Cevaxin
Locations (3):
- Panama (3):
  - Cevaxin - 24 de Diciembre, Panama City
  - Cevaxin - Chorrera, Panama City
  - Cevaxin-- Avenida Mexico, Panama City

IPD SHARING:
Plan to Share IPD: No